CLINICAL TRIAL: NCT02446561
Title: A Study of Whether 3 New Oral Formulations of a Strong Pain Killer Release the Same Amount of Drug Into the Body as the Marketed Medication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HMX1509
Record Dates: First submitted 2015-04-22; First posted 2015-05-18 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Pain
Keywords: Healthy Volunteer; Pharmacokinetics
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MRXXX (Active Comparator): Active comparator
  Interventions: Drug: MRXXX
- MR1XXX (Experimental): MR1XXX
  Interventions: Drug: MR1XXX
- MR2XXX (Experimental): MR2XXX
  Interventions: Drug: MR2XXX
- MR3XXX (Experimental): MR3XXX
  Interventions: Drug: MR3XXX

INTERVENTIONS:
Drug: MRXXX
  Arms: MRXXX
Drug: MR1XXX
  Arms: MR1XXX
Drug: MR2XXX
  Arms: MR2XXX
Drug: MR3XXX
  Arms: MR3XXX

SUMMARY:
To determine whether three new oral formulations of a strong pain killer release the drug into the body in a similar pattern as the already marketed reference capsule formulation with or without food

DETAILED DESCRIPTION:
Comparisons will be made between three new oral formulations and an existing marketed reference capsule formulation to determine whether the release rates of the products are similar or equivalent in a fed or fasted state. Determination is by measurement of drug concentrations in the blood at serial collection time points pre-dose until 72 hours post-dose, following an administration of a single oral dose. Pharmacokinetics parameters of AUC and Cmax are the primary endpoints

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Healthy male or female subjects aged 18 to 55 inclusive.
3. Female subjects of child bearing potential must be willing to use two highly effective methods of contraception throughout the study, one of which must include a barrier method.
4. Female subjects who are post-menopausal (defined as spontaneous amenorrhea for at least a year) or permanently sterilised (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy). These subjects are not required to use any contraception.
5. Male subjects must be willing to use contraception with their partners throughout the study and for 30 days after completion of the study and agree to inform the Investigator if their partner becomes pregnant during this time.
6. Body weight ranging from 55 to 100 kg and a BMI ≥ 18.5 and ≤ 30.0.
7. Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
8. Willing to eat all the food supplied throughout the study.
9. The subject's primary care physician has confirmed within the last 12 months of first dosing that there is nothing in their medical history that would preclude their enrolment into a clinical study

Exclusion Criteria:

1. Any history of drug or alcohol abuse.
2. Any history of conditions that might interfere with drug absorption, distribution, metabolism or excretion.
3. Use of opioid or opioid antagonist-containing medication in the past 30 days.
4. Any history of frequent nausea or vomiting regardless of etiology.
5. Any history of seizures or symptomatic head trauma.
6. Any history of paralytic ileus, respiratory depression, hypoxia or elevated carbon dioxide levels in the blood.
7. Participation in a clinical drug study during the 90 days preceding the initial dose in this study.
8. Subjects must not participate in both the pilot phase and the definitive phase of the study, or in more than one Cohort.
9. Any significant illness during the 4 weeks preceding entry into this study.
10. Use of any medication including vitamins, herbal and/or mineral supplements during the 7 days preceding the initial dose or during the course of this study (with the exception of the continued use of HRT and contraceptives).
11. Refusal to abstain from food 8 hours preceding and 4 hours following study drug administration, to abstain from foods containing poppy seeds 48 hours preceding and entirely during each confinement, and to abstain from caffeine or xanthine containing food or beverages and grapefruit juice within 48 hours before IMP administration and for the duration of study confinement until after the last study PK sample has been taken in each study period.
12. Weekly alcohol intake exceeding the equivalent of 14 units/week for females and 21 units/week for males. (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
13. Consumption of alcoholic beverages within 48 hours before study drug administration, and refusal to abstain from alcohol for the duration of the study confinement and for at least 48 hours after the last naltrexone dose in each study period.
14. History of smoking within 45 days of study drug administration and refusal to abstain from smoking during the study.
15. Blood or blood products donated within 90 days prior to study drug administration or any time during the study, except as required by this protocol.
16. Positive results of urine drug screen, alcohol test, pregnancy test, HBsAg, Hepatitis C antibody, or HIV tests.
17. Refusal to allow their primary care physician to be informed of participation in the trial.
18. Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence as measured by PK parameters | Up to 72 hours
  AUCt, AUCINF, LambdaZ, t1/2Z, Cmax and tmax

SECONDARY OUTCOMES:
Safety and tolerability as measured by adverse events, vital signs, clinical lab results and ECGs. | Up to 7-10 days after last dose
  Collection of adverse events, vital signs, clinical lab results and ECGs.

CONTACTS AND LOCATIONS:
Locations (1):
- BioKinetic Europe Ltd, Belfast, United Kingdom